CLINICAL TRIAL: NCT04819581
Title: An Open-label, Randomized, Four-treatment, Four-sequence, Four-period, Crossover, Pharmacokinetic Study of SP-103 in Healthy Adult Human Subjects
Brief Title: Pharmacokinetic Study of SP-103 in Healthy Adult Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scilex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCI-LIDO-PK-005
Record Dates: First submitted 2021-03-23; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SP-103 (1 topical system) (Experimental): One topical system applied to the skin on the back for 12 hours.
  Interventions: Drug: SP-103
- SP-103 (2 topical systems) (Experimental): Two topical systems applied to the skin on the back for 12 hours.
  Interventions: Drug: SP-103
- SP-103 (3 topical systems) (Experimental): Three topical systems applied to the skin on the back for 12 hours.
  Interventions: Drug: SP-103
- ZTlido (Active Comparator): Three topical systems applied to the skin on the back for 12 hours.
  Interventions: Drug: ZTlido

INTERVENTIONS:
Drug: SP-103 — lidocaine topical system 5.4%
  Arms: SP-103 (1 topical system); SP-103 (2 topical systems); SP-103 (3 topical systems)
Drug: ZTlido — lidocaine topical system 1.8%
  Arms: ZTlido

SUMMARY:
This study will assess the systemic exposure and pharmacokinetic parameters of SP-103 topical system following one, two, or three topical system applications and compare to the pharmacokinetics of ZTlido.

ELIGIBILITY:
Key Inclusion Criteria:

* Must be healthy based on by medical history, laboratory work, ECG, and physical exam
* Body mass index ranging between 18.0-32.5 kg/m2, inclusive
* If childbearing potential, use of acceptable form of birth control
* In the case of females of childbearing potential, have a negative serum pregnancy test

Key Exclusion Criteria:

* Allergy or known hypersensitivity to lidocaine, amide-type local anesthetics or any component of the product formulation
* Any major medical illness 3 months prior or any significant history or ongoing chronic medical illness affecting the major body systems, including the skin
* Subjects with conditions that might affect application of the product or its adhesive properties (including psoriasis, eczema, atopic dermatitis, damaged or irritated epidermal layer, and excessive hair or oil on the skin)
* Use of antiarrhymthic drugs (such as tocainide and mexiletine) and local anesthetics within 14 days prior to product application.
* History of addiction, abuse, or misuse of any drug
* Use of nicotine-containing products within 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-08-03 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of lidocaine | 0, 2, 4, 6, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22, 24, 48 hours post-dose
  Peak plasma concentration of lidocaine after 12 hour topical system application
Area under the Plasma-Concentration Time Curve (AUC) from Time 0 to Time 48 hours | 0, 2, 4, 6, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22, 24, 48 hours post-dose
  Area under the plasma concentration versus time curve from 0 to 48 hours of lidocaine in plasma
Area under the Plasma-Concentration Time Curve (AUC) from Time 0 to Time Infinity | 0, 2, 4, 6, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22, 24, 48 hours post-dose
  Area under the plasma concentration versus time curve from 0 to infinite time of lidocaine in plasma

SECONDARY OUTCOMES:
Mean adhesion score | 0, 3, 6, 9, 12 hours post-dose
  Adhesion to skin assessed by FDA 0-4 scoring system. The scoring for adhesion of patches is indicated as follows: 0 = ≥ 90% Adhered (essentially no lift off the skin), 1 = ≥ 75% to < 90% Adhered (some edges only lifting off the skin), 2 = ≥ 50% to < 75% Adhered (less than half of the patch lifting off the skin), > 0% to < 50% Adhered but not detached (more than half of the patch lifting off the skin without falling off), and 4 = 0% adhered (patched completely detached). The mean score is calculated as the average of scores at time 3, 6, 9, and 12 hours.
Dermal response score | 12.5 and 14 hours post-dose
  Product tolerability is assessed by Dermal Response Score. The application site is evaluated 30 minutes and 2 hours after product removal (12.5 and 14 hours post-dose, respectively). Response score from 0 to 7; 0= No evidence of irritation, 1= Minimal erythema, barely perceptible, 2= Definite erythema, readily visible; minimal edema or minimal papular response, 3= Erythema and papules, 4= Definite edema, 5= Erythema, edema and papules, 6= Vesicular eruption, 7= Strong reaction spreading beyond test (i.e., application) site.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Boldingh, PharmD, Principal Investigator — AXIS Clinicals
Locations (1):
- AXIS Clinicals, Dilworth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No